CLINICAL TRIAL: NCT06672237
Title: MAGNITUDE-2: A Phase 3, Multinational, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of NTLA-2001 in Participants With Hereditary Transthyretin Amyloidosis With Polyneuropathy (ATTRv-PN)
Brief Title: A Phase 3 Study of NTLA-2001 in ATTRv-PN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intellia Therapeutics (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITL-2001-CL-311
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Neuromuscular Disease; Neuromuscular Diseases (NMD); Neurodegenerative Disease; Neurodegenerative Disease, Hereditary; Neurodegenerative Diseases; Neuromuscular Diseases; Nerve Disorders; Nervous System Disease; Nervous System Diseases; Genetic Disease, Inborn; Amyloidosis, Familial; Amyloidosis, Hereditary; Amyloidosis; Polyneuropathies; Amyloid Neuropathies; Amyloid Neuropathies, Familial; Peripheral Nervous System Disease; Peripheral Nervous System Diseases; Metabolism, Inborn Errors; Metabolic Diseases
Keywords: TTR; Amyloidosis; Polyneuropathy; NTLA-2001; ATTR; ATTR-PN; ATTRv-PN; Transthyretin; TTR-mediated amyloidosis; Amyloidosis, hereditary; Amyloidosis, hereditary, transthyretin-related amyloidosis; Transthretin amyloid polyneuropathy; TTR PN; TTR polyneuropathy; nexiguran ziclumeran; nex-z
MeSH Terms: conditions — Neuromuscular Diseases; Neurodegenerative Diseases; Heredodegenerative Disorders, Nervous System; Nervous System Diseases; Genetic Diseases, Inborn; Amyloidosis, Familial; Amyloidosis; Polyneuropathies; Amyloid Neuropathies; Amyloid Neuropathies, Familial; Peripheral Nervous System Diseases; Metabolism, Inborn Errors; Metabolic Diseases; Amyloidosis, Hereditary, Transthyretin-Related | interventions — NTLA-2001; Saline Solution

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in a 1:1 ratio to nexiguran ziclumeran or placebo with opportunity for crossover.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- nexiguran ziclumeran (Experimental): nexiguran ziclumeran 55 mg by single IV infusion
  Interventions: Biological: nexiguran ziclumeran
- Normal Saline (Placebo Comparator): Placebo; Normal saline (0.9% NaCl) by single IV infusion
  Interventions: Drug: Normal Saline as Placebo

INTERVENTIONS:
Biological: nexiguran ziclumeran — nexiguran ziclumeran 55 mg by single IV infusion
  Other Names: NTLA-2001
  Arms: nexiguran ziclumeran
Drug: Normal Saline as Placebo — Normal saline (0.9% NaCl) by single IV infusion
  Arms: Normal Saline

SUMMARY:
This study will be conducted to evaluate the efficacy and safety of a single dose of nexiguran ziclumeran (NTLA-2001) compared to placebo in participants with ATTRv-PN.

DETAILED DESCRIPTION:
This is a multinational, multicenter, double-blind, placebo-controlled study in approximately 50 participants, who will be randomized 1:1 to receive a single infusion of either nexiguran ziclumeran or placebo. To ensure all participants will have the potential to receive nexiguran ziclumeran, participants will have the option to cross over to the opposite study arm at Month 12 or Month 18, depending on study criteria.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ATTRv-PN
* Karnofsky Performance Status (KPS) ≥ 60

Exclusion Criteria:

* Other causes of amyloidosis (amyloidosis caused by non-TTR protein)
* Other known causes of sensorimotor or autonomic neuropathy
* Diabetes mellitus
* New York Heart Association Class III or IV heart failure
* Liver failure
* Hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection
* Prior receipt of a TTR silencer (Small interfering RNA (siRNA) or Antisense oligonucleotides (ASOs))
* Estimated Glomerular Filtration Rate < 30 mL/min/1.73 m2
* Unable or unwilling to take vitamin A supplementation for the duration of the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Modified Neuropathy Impairment Score +7 (mNIS+7) | 18 Months
Serum TTR | 29 Days

SECONDARY OUTCOMES:
Norfolk Quality of Life-Diabetic Neuropathy (Norfolk QoL-DN) Questionnaire | 18 Months
Modified Body Mass Index (mBMI) | 18 Months
Serum TTR | 18 Months

CONTACTS AND LOCATIONS:
Locations (16):
- Argentina (3):
  - Hospital Británico de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires (HIBA), Buenos Aires
  - Hospital El Cruce, San Juan Bautista
- Westmead Hospital, Westmead, Australia
- Brazil (4):
  - Hospital das Clinicas da Universidade Estadual de Campinas (UNICAMP), Campinas
  - HCFMRP - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto, Ribeirão Preto
  - Instituto de Educacao, Pesquisa e Gestao em Saude, Rio de Janeiro
  - PSEG Centro de Pesquisa Clinica S.A., São Paulo
- National Institute of Medical Sciences and Nutrition - Salvador Zubiran (INCMNSZ), Tlalpan, Mexico
- New Zealand Clinical Research, Auckland, New Zealand
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation - Linkou Branch, Taoyuan District
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No